CLINICAL TRIAL: NCT07238920
Title: Closed-Loop Neurofeedback Targeting the Right Dorsolateral Prefrontal Cortex for Cardiac Autonomic Modulation in Coronary Artery Disease With Anxiety - A Randomized, Sham-Controlled Trial
Brief Title: Closed-Loop Neurofeedback Targeting the Right Dorsolateral Prefrontal Cortex for Cardiac Autonomic Modulation in Coronary Artery Disease With Anxiety
Acronym: HEART-SET-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Medical College (Other)
Collaborators: The Second Hospital of Shenyang Medical College (Other)
Responsible Party: Principal Investigator, Lin Tao, Assoc.Prof., Shenyang Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEART-SET-1
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Coronary Heart Disease (CHD); Anxiety Disorders
Keywords: Coronary heart disease; Anxiety; Neurofeedback; Heart rate variability
MeSH Terms: conditions — Coronary Disease; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study adopts a parallel-group, randomised, sham-controlled design to investigate whether real-time fNIRS-based neurofeedback targeting the right dorsolateral prefrontal cortex (right DLPFC) can modulate cardiac autonomic function in patients with stable coronary heart disease (CHD) and comorbid anxiety. Participants are randomly assigned (1:1) to either the real neurofeedback group or the sham feedback group. Both groups receive visual feedback derived from their own right DLPFC activation data during an identical auditory stimulation paradigm (1 Hz amplitude-modulated pure tone at ~60 dB with randomly embedded 10-second white noise segments), while fNIRS and ECG are recorded simultaneously.
Who Masked: Participant, Outcomes Assessor
Masking Description: Real Neurofeedback Group Participants receive real-time visual feedback based on activation of the right dorsolateral prefrontal cortex (right DLPFC), computed with a stringent statistical threshold (T = -3.3). This threshold enables high-sensitivity coupling between neural activity and the energy bar displayed on screen. The interface omits numerical values, and participants are blinded to both group allocation and threshold settings, ensuring a causally interpretable closed-loop training.
  Sham Neurofeedback Group Participants receive feedback using a lenient threshold (T = -1), greatly reducing the effective coupling between right DLPFC activation and the visual feedback. The screen interface is identical to the real group, and no numerical values are shown. Participants are blinded to their group and threshold settings, limiting the possibility of meaningful self-regulation.
  Both groups undergo identical auditory stimulation paradigms, noise overlay protocols, and testing procedures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Neurofeedback Group (Experimental): Participants receive real-time visual feedback based on activation of the right dorsolateral prefrontal cortex (right DLPFC), computed with a stringent statistical threshold (T = -3.3). This threshold enables high-sensitivity coupling between neural activity and the energy bar displayed on screen. The interface omits numerical values, and participants are blinded to both group allocation and threshold settings, ensuring a causally interpretable closed-loop training.
  Interventions: Device: Real-time fNIRS-ECG neurofeedback
- Sham Neurofeedback Group (Sham Comparator): Participants receive feedback using a lenient threshold (T = -1), greatly reducing the effective coupling between right DLPFC activation and the visual feedback. The screen interface is identical to the real group, and no numerical values are shown. Participants are blinded to their group and threshold settings, limiting the possibility of meaningful self-regulation.
  Interventions: Device: Real-time fNIRS-ECG neurofeedback

INTERVENTIONS:
Device: Real-time fNIRS-ECG neurofeedback — This intervention uses real-time neurofeedback based on right dorsolateral prefrontal cortex (right DLPFC) activity measured by functional near-infrared spectroscopy (fNIRS), with simultaneous ECG recording. During a slow-wave auditory paradigm (1 Hz amplitude-modulated tone with embedded white noise), participants attempt to downregulate right DLPFC activation via active volitional strategies, guided by a visual energy bar.
  Before formal intervention, a 3-day adaptation phase familiarises participants with the interface and task, under guidance. The formal training occurs on Days 4-5 (15 blocks/day), using identical auditory input and recording protocol. Participants are randomised to real or sham feedback groups, differing only in the statistical threshold used to generate feedback (T = -3.3 vs T = -1.0). Participants and assessors are blinded to allocation.

SUMMARY:
The goal of this clinical trial is to test whether real-time fNIRS-BCI neurofeedback targeting the right dorsolateral prefrontal cortex (right DLPFC), using active volitional control during a slow-wave auditory acoustic paradigm, can suppress cardiac sympathetic activity and improve autonomic regulation in right-handed patients with stable coronary heart disease (CHD) and comorbid DSM-5 anxiety.

The main questions it aims to answer are:

Does real neurofeedback, compared with sham, reduce baseline-corrected heart rate during the auditory stimulation window? Does real neurofeedback, compared with sham, increase HRV spectral power around 0.0167 Hz (1/60 Hz) and produce stronger suppression of right DLPFC activation? Does suppression of right DLPFC activation mediate the effect of group assignment on heart rate?

If there is a comparison group: Researchers will compare the real neurofeedback group with the sham (non-contingent) feedback group, which uses identical audio and interface, to determine whether coupling feedback to right DLPFC activity yields autonomic benefits.

Participants will:

Complete eligibility screening in cardiology and psychiatry and provide informed consent; baseline demographics, medical history, vital signs, and medications are recorded (HAMA/HAMD used for eligibility only).

Undergo a 3-day adaptation phase to practice active volitional self-regulation while viewing a real-time energy bar mapped to right DLPFC statistics; adaptation data are not analyzed for outcomes.

Attend two formal sessions (Days 4-5), each with 15 blocks of 60 s (20 s rest + 40 s stimulus). The auditory stimulus is a 1 Hz amplitude-modulated pure tone at approximately 60 dB; 10-second white-noise bursts are randomly embedded within the 40-second window. During the stimulation period, participants receive real or sham feedback on right DLPFC activation and act to push the energy bar below an unlabeled threshold line using active volitional strategies.

Undergo synchronous fNIRS (HbO) and 3-lead ECG (1,000 Hz) recording throughout; online processing and rendering performance metrics are logged; adverse events are monitored and managed per protocol.

DETAILED DESCRIPTION:
This study is a randomised, sham-controlled, parallel-group neurofeedback trial designed to test whether real-time fNIRS-BCI targeting the right dorsolateral prefrontal cortex (right DLPFC), using active volitional control during a slow-wave auditory acoustic paradigm, can suppress cardiac sympathetic activity and improve autonomic regulation in right-handed patients with stable coronary heart disease and comorbid DSM-5 anxiety. Eligibility criteria, outcome measures, arms and interventions, and statistical analysis are specified in their dedicated fields of this record to avoid duplication.

Participants complete screening and a three-day adaptation phase, followed by two formal experimental sessions on consecutive days. No verbal guidance is provided on test days. During each formal session, participants undergo 15 block cycles of 60 seconds each, comprising 20 seconds of rest and 40 seconds of auditory stimulation. The auditory stimulus is a 1 Hz amplitude-modulated pure tone at approximately 60 dB. Within the 40-second window, a 10-second white-noise burst is randomly embedded while avoiding the first and last 2 seconds; start times are selected without replacement from a discrete set to minimise predictability and sequence effects and to probe interference resistance.

Neurofeedback targets the right DLPFC. Real-time statistical values of cortical activation are mapped to a visual energy bar that serves as the feedback signal. Participants use active volitional strategies to push the energy bar below an unlabeled threshold line during stimulation. In the real-feedback group the statistical threshold is set to T = -3.3, producing a sensitive, contingent mapping between right DLPFC activity and the energy bar. In the sham-feedback group the threshold is set to T = -1, weakening the effective coupling between neural state and on-screen feedback while keeping the interface identical. Only the session operator is aware of group assignment; outcome assessors and data analysts are blinded.

Signals are acquired synchronously. fNIRS uses a NirSmart system with 7 sources and 7 detectors forming 19 channels, dual wavelengths at 730 nm and 850 nm, source-detector separation of 3 cm, and an 11 Hz sampling rate with avalanche photodiode detectors. Optodes are positioned over bilateral prefrontal cortex using the 10-20 system with FPz as the central reference. Channels are co-registered to MNI space, with right DLPFC (Brodmann area 46) designated a priori as the region of interest; channels 11 and 13 represent right DLPFC for feedback, and channels 17 and 18 represent left DLPFC for reference. ECG is recorded using a 3-lead configuration at 1,000 Hz.

Online processing and feedback are implemented with the NeuroMind-NIRS pipeline. A MATLAB timer provides a fixed update cadence. The streaming architecture is layered into data, visualisation, control, and persistence channels. A sliding-window general linear model is applied to fNIRS signals with low-pass filtering, linear detrending, and within-window normalisation. A boxcar task regressor convolved with a canonical haemodynamic response function is used; the statistical readout at the end of each window updates the energy bar and threshold decision. Statistical inference is prioritised ahead of rendering within a fixed real-time budget to maintain a stable feedback cadence. Per-frame compute time, render time, total pipeline time, latency, and dropped-frame rate are logged. The acoustic stimulus is not triggered or gated by the statistical readout.

Offline fNIRS preprocessing is performed in MATLAB using the Homer2 toolbox. Steps include conversion to optical density, motion artefact detection by channel, spline interpolation correction, band-pass filtering at 0.01 to 0.08 Hz, and calculation of oxyhaemoglobin concentration via the modified Beer-Lambert law. Analyses focus on HbO due to its higher signal-to-noise ratio. For activation analysis, normalised HbO time series from DLPFC channels enter a general linear model with a task regressor based on the convolved canonical haemodynamic response function and its derivatives; preprocessed ECG-derived covariates are included to account for low-frequency physiological oscillations. Subject-level task β estimates are taken forward to group-level linear mixed-effects models.

ECG processing includes R-peak detection by the Pan-Tompkins algorithm, correction of spurious detections, construction of RR interval series, ectopic beat removal using robust filters, and resampling as needed for alignment with fNIRS. Heart rate and heart rate variability are computed within block-aligned windows with baseline correction using the pre-stimulation interval. For spectral analysis, time-frequency methods are applied to quantify power around 0.0167 Hz, corresponding to the 60-second block rhythm within the very low frequency band.

Safety is monitored continuously from the start of adaptation through the end of Session 2. Anticipated adverse events related to sympathetic attenuation include mild dizziness or drowsiness, transient bradycardia or hypotension-related discomfort, headache, and nausea. Standard operating procedures specify pausing or terminating sessions and initiating clinical assessment as needed; serious adverse events trigger immediate discontinuation and follow-up. Quality control includes unscheduled supervisory checks, standardised operator training, checkpointed critical steps, real-time records, de-identified data handling, tiered access control, and auditable transfer logs. De-identified individual data and analysis scripts will be shared on a recognised repository at publication in accordance with data use and ethics policies.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years, any sex.
* Right-handed, with resting heart rate between 60 and 100 beats per minute.
* Confirmed diagnosis of CHD, defined as at least one of the following:

  (i) positive stress test; (ii) documented myocardial infarction (MI) with electrocardiographic changes and concurrent elevation of creatine kinase MB isoenzyme or troponin; (iii) angiographically confirmed coronary atherosclerosis with ≥50% stenosis in at least one coronary artery.
* Diagnosis of an anxiety disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
* Hamilton Anxiety Rating Scale (HAMA) score ≥16 and 17-item Hamilton Depression Rating Scale (HAMD-17) score ≤17.

Exclusion Criteria:

* Acute unstable angina.
* Severe congestive heart failure (New York Heart Association [NYHA] class IV).
* Valvular heart disease.
* History of atrial fibrillation.
* Unstable blood pressure, defined as systolic blood pressure >180 mmHg or <90 mmHg.
* Pregnancy.
* History of unstable medical conditions, including cerebrovascular disease, dementia, hyperthyroidism, pulmonary disease, or malignancy. These are assessed through medical history, electronic health records, physical examination, and ECG findings.
* High risk of suicide or homicide.
* Presence of other psychiatric disorders, including psychotic disorders, bipolar disorder, or active substance use disorders.
* Use of psychotropic medication within 1 month prior to enrolment, to avoid potential interference with haemodynamic measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
The between-group difference (real neurofeedback vs sham) in baseline-corrected heart rate (HR) during the task stimulation window. | The formal experimental phase (day 4 and 5).

SECONDARY OUTCOMES:
Between-group difference in task-related activation of the right dorsolateral prefrontal cortex (right DLPFC). | The formal experimental phase (day 4 and 5).
  Quantified as the GLM task regressor β (HbO) during the slow-wave auditory neurofeedback paradigm
Between-group difference in HRV spectral power at 0.0167 Hz during the task stimulation window, based on wavelet time-frequency analysis. | The formal experimental phase (day 4 and 5).

OTHER OUTCOMES:
Mediation analysis: to assess the indirect effect of group assignment on baseline-corrected HR via changes in right DLPFC activation. | The formal experimental phase (day 4 and 5).
Incidence of any adverse events during training or stimulation (e.g., mild dizziness or drowsiness, transient bradycardia or blood pressure-related discomfort, headache, or nausea). | From the adaptation phase until completion of the formal experimental sessions (Days 1-5).

CONTACTS AND LOCATIONS:
Overall Officials: Yun-En Liu, MD, Study Chair — Shenyang Medical College; Lin Tao, MM, Principal Investigator — Shenyang Medical College

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, study protocol, MATLAB scripts, and supporting materials will be made publicly available at the time of formal publication. Data will be hosted on an internationally recognised third-party repository and accessible for non-commercial scientific use.
Supporting Information: Study Protocol
Time Frame: available at the time of formal publication